CLINICAL TRIAL: NCT02548689
Title: Evaluating PAI-1 Expression in the Hair Follicles of Patients With Non-scarring Hair Loss.
Brief Title: PAI-1 Expression in Non-scarring Hair Loss
Status: Terminated | Type: Observational
Why Stopped: Original lead investigator left Northwestern University
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Maria Colavincenzo, Assistant Professor in Dermatology, Northwestern University
Other Study IDs: STU00103009
Record Dates: First submitted 2015-08-03; First posted 2015-09-14 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Androgenetic Alopecia; Telogen Effluvium; Alopecia Areata
Keywords: alopecia; hair loss
MeSH Terms: conditions — Alopecia; Alopecia Areata

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin tissue will be formalin-fixed overnight at room temperature, processed and paraffin embedded. Six micron thick sections will be prepared. Tissue blocks and slides will be stored at room temperature. All samples will be de-identified.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-scarring hair loss: Patients seen at Northwestern Memorial Hospital or Northwestern Medical Faculty Foundation physician offices that have undergone evaluation for hair loss and have a diagnosis of androgenetic alopecia, telogen effluvium or alopecia areata.
- Control: Age-matched controls who do not have a history of hair loss and have normal scalp skin without evidence of hair loss.

SUMMARY:
This study will investigate whether subjects who suffer from hair loss have increased levels of PAI-1 compared to age-matched control subjects. The level of PAI-1 expression will be determined in subjects without hair loss and in subjects with non-scarring hair loss, including androgenetic alopecia, telogen effluvium and alopecia areata.

DETAILED DESCRIPTION:
This study will compare the levels of PAI-1 expression in subjects with different forms of non-scarring hair loss and in these subjects vs normal age-matched controls. Hair loss subjects will have their Northwestern Memorial Hospital and Northwestern Medical Faculty Foundation medical records reviewed to ensure they meet inclusion and exclusion criteria. All subjects will have a 4 mm punch biopsy on the scalp. Tissue PAI-1 levels from scalp skin biopsies will be determined by immunohistochemical staining. Samples will be kept for approximately 15 years, after which time unused samples will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Age-matched control subjects who do not have a history of hair loss
* A clinical and pathologic diagnosis of androgenetic alopecia, telogen effluvium, alopecia areata or normal scalp skin
* All subjects must have given signed, informed consent prior to registration in study

Exclusion Criteria:

* History of previous hair transplantation
* Current and past use of medications topically on the scalp
* Clinical or pathologic diagnosis of a scarring alopecia
* History of inflammatory conditions of the scalp such as psoriasis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All hair loss subjects will be recruited from patients seen at Northwestern Memorial Hospital or Northwestern Medical Faculty Foundation physicians offices. Age-matched control subjects will be recruited by either 1) the use of flyers displayed in the hospital and surrounding community, or 2) will be identified during a clinic visit at Northwestern Memorial Hospital or Northwestern Medical Faculty Foundation physician offices.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
PAI-1 expression level in scalp skin biopsy samples | Baseline
  Tissue PAI-1 expression levels will be determined by immunohistochemistry, a three-layer biotin-strepavidin system. Positive PAI-1 expression per total tissue area will be quantified using the color-picker function in imaging software.The PAI-1 expression found in normal scalps will be compared to those found in scalps with hair loss.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Colavincenzo, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Norwood OT. Incidence of female androgenetic alopecia (female pattern alopecia). Dermatol Surg. 2001 Jan;27(1):53-4. PMID 11231244
- [Background] Scheinfeld N. A review of hormonal therapy for female pattern (androgenic) alopecia. Dermatol Online J. 2008 Mar 15;14(3):1. PMID 18627703
- [Background] Cash TF. The psychological effects of androgenetic alopecia in men. J Am Acad Dermatol. 1992 Jun;26(6):926-31. doi: 10.1016/0190-9622(92)70134-2. PMID 1607410
- [Background] Cash TF, Price VH, Savin RC. Psychological effects of androgenetic alopecia on women: comparisons with balding men and with female control subjects. J Am Acad Dermatol. 1993 Oct;29(4):568-75. doi: 10.1016/0190-9622(93)70223-g. PMID 8408792
- [Background] Ogunmakin KO, Rashid RM. Alopecia: the case for medical necessity. Skinmed. 2011 Mar-Apr;9(2):79-84. PMID 21548511
- [Background] Rogers NE, Avram MR. Medical treatments for male and female pattern hair loss. J Am Acad Dermatol. 2008 Oct;59(4):547-66; quiz 567-8. doi: 10.1016/j.jaad.2008.07.001. PMID 18793935
- [Background] Mounsey AL, Reed SW. Diagnosing and treating hair loss. Am Fam Physician. 2009 Aug 15;80(4):356-62. PMID 19678603
- [Background] Rathnayake D, Sinclair R. Male androgenetic alopecia. Expert Opin Pharmacother. 2010 Jun;11(8):1295-304. doi: 10.1517/14656561003752730. PMID 20426708
- [Background] Rossi A, Cantisani C, Melis L, Iorio A, Scali E, Calvieri S. Minoxidil use in dermatology, side effects and recent patents. Recent Pat Inflamm Allergy Drug Discov. 2012 May;6(2):130-6. doi: 10.2174/187221312800166859. PMID 22409453
- [Background] Schweiger ES, Boychenko O, Bernstein RM. Update on the pathogenesis, genetics and medical treatment of patterned hair loss. J Drugs Dermatol. 2010 Nov;9(11):1412-9. PMID 21061765
- [Background] Mella JM, Perret MC, Manzotti M, Catalano HN, Guyatt G. Efficacy and safety of finasteride therapy for androgenetic alopecia: a systematic review. Arch Dermatol. 2010 Oct;146(10):1141-50. doi: 10.1001/archdermatol.2010.256. PMID 20956649
- [Background] Berkenpas MB, Lawrence DA, Ginsburg D. Molecular evolution of plasminogen activator inhibitor-1 functional stability. EMBO J. 1995 Jul 3;14(13):2969-77. doi: 10.1002/j.1460-2075.1995.tb07299.x. PMID 7621813
- [Background] Eren M, Gleaves LA, Atkinson JB, King LE, Declerck PJ, Vaughan DE. Reactive site-dependent phenotypic alterations in plasminogen activator inhibitor-1 transgenic mice. J Thromb Haemost. 2007 Jul;5(7):1500-8. doi: 10.1111/j.1538-7836.2007.02587.x. Epub 2007 Apr 16. PMID 17439629
- [Background] Bahta AW, Farjo N, Farjo B, Philpott MP. Premature senescence of balding dermal papilla cells in vitro is associated with p16(INK4a) expression. J Invest Dermatol. 2008 May;128(5):1088-94. doi: 10.1038/sj.jid.5701147. Epub 2007 Nov 8. PMID 17989730
- [Background] Simonetti O, Lucarini G, Bernardini ML, Simoncini C, Biagini G, Offidani A. Expression of vascular endothelial growth factor, apoptosis inhibitors (survivin and p16) and CCL27 in alopecia areata before and after diphencyprone treatment: an immunohistochemical study. Br J Dermatol. 2004 May;150(5):940-8. doi: 10.1111/j.1365-2133.2004.05881.x. PMID 15149507
- [Background] Trueb RM. Oxidative stress in ageing of hair. Int J Trichology. 2009 Jan;1(1):6-14. doi: 10.4103/0974-7753.51923. PMID 20805969
- [Background] Balsara RD, Castellino FJ, Ploplis VA. A novel function of plasminogen activator inhibitor-1 in modulation of the AKT pathway in wild-type and plasminogen activator inhibitor-1-deficient endothelial cells. J Biol Chem. 2006 Aug 11;281(32):22527-36. doi: 10.1074/jbc.M512819200. Epub 2006 Jun 19. PMID 16785241
- [Background] Kortlever RM, Higgins PJ, Bernards R. Plasminogen activator inhibitor-1 is a critical downstream target of p53 in the induction of replicative senescence. Nat Cell Biol. 2006 Aug;8(8):877-84. doi: 10.1038/ncb1448. Epub 2006 Jul 23. PMID 16862142
- [Background] Ploplis VA, Balsara R, Sandoval-Cooper MJ, Yin ZJ, Batten J, Modi N, Gadoua D, Donahue D, Martin JA, Castellino FJ. Enhanced in vitro proliferation of aortic endothelial cells from plasminogen activator inhibitor-1-deficient mice. J Biol Chem. 2004 Feb 13;279(7):6143-51. doi: 10.1074/jbc.M307297200. Epub 2003 Nov 18. PMID 14625301
- [Background] Takeshita K, Yamamoto K, Ito M, Kondo T, Matsushita T, Hirai M, Kojima T, Nishimura M, Nabeshima Y, Loskutoff DJ, Saito H, Murohara T. Increased expression of plasminogen activator inhibitor-1 with fibrin deposition in a murine model of aging, "Klotho" mouse. Semin Thromb Hemost. 2002 Dec;28(6):545-54. doi: 10.1055/s-2002-36699. PMID 12536348
- [Background] Vaughan DE. PAI-1 antagonists: the promise and the peril. Trans Am Clin Climatol Assoc. 2011;122:312-25. PMID 21686234
- [Background] Vaughan DE, De Taeye BM, Eren M. PAI-1 antagonists: predictable indications and unconventional applications. Curr Drug Targets. 2007 Sep;8(9):962-70. doi: 10.2174/138945007781662364. PMID 17896947
- [Background] Angleton P, Chandler WL, Schmer G. Diurnal variation of tissue-type plasminogen activator and its rapid inhibitor (PAI-1). Circulation. 1989 Jan;79(1):101-6. doi: 10.1161/01.cir.79.1.101. PMID 2491971